CLINICAL TRIAL: NCT00553917
Title: Study of the Pharmacokinetics and Pharmacogenetics of Selective Serotonin Reuptake Inhibitors During Pregnancy
Brief Title: Study to Evaluate the Effectiveness of Certain Selective Serotonin Reuptake Inhibitor (SSRI) Antidepressants During Pregnancy and Evaluate Newborn Outcomes
Status: Terminated | Type: Observational
Why Stopped: Poor recruitment to experimental arms and study remained unfunded
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 0708-10
Record Dates: First submitted 2007-11-05; First posted 2007-11-06 (Estimated); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Depression
Keywords: Pregnancy; Depression; Antidepressants
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole Blood Plasma human milk
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1: Pregnant women currently taking Prozac for the treatment of depression
- 2: Pregnant women currently taking Zoloft for the treatment of depression
- 3: Pregnant women not currently using medication for the treatment of depression
- 4: Pregnant women with no history of, symptoms of, or treatment for depression

SUMMARY:
The purpose of this study is to evaluate if during pregnancy, a common group of antidepressant medications (SSRI's) adequately treats the symptoms of depression and to evaluate if there are any effects of these medications on the newborn infant.

DETAILED DESCRIPTION:
The amount or levels of some antidepressant medications in the blood (e.g. selective serotonin reuptake inhibitors or SSRIs) seem to be decreased during pregnancy. If the levels of SSRIs in the blood are low, the medication may not be adequately treating depression. The objective of our study is to evaluate whether pregnant women have decreased levels of SSRIs and a resultant decreased improvement of depression with SSRIs. We also want to evaluate whether variations in the genes related to how the body eliminates the SSRIs or how the SSRIs work influence the improvement in the depression pregnant women experience from these drugs. We will conduct a study in 100 pregnant women who are receiving fluoxetine (n = 25) or sertraline (n = 25) for the treatment of depression, who are not receiving any medication for depression (n = 25), or who are pregnant no history or treatment for depression (n= 25). Participants will be enrolled any time before 26 weeks of pregnancy. Blood samples will be collected for genetic analysis in all subjects, and for drug level measurements during pregnancy, at delivery, and post partum in the subjects taking antidepressant medication. We will also be monitoring monthly platelet serotonin levels in all groups. In addition, the scores of a rating scale to measure the severity of depression and two rating scales to measure the undesirable effects of the treatment will be obtained on enrollment and monthly for up to 12 weeks after delivery. Maternal and umbilical cord blood samples will be obtained at delivery for determination of SSRI levels, platelet serotonin levels (a marker that SSRIs are working), and for collection of neonatal DNA. After delivery all mothers will complete a survey about how she is feeling about herself and the baby, and the baby's behavior will be observed for a 1 hour time interval. Babies of mothers taking medication will have a blood sample drawn at 2-3 months after birth to measure the drug level as compared with cord blood sample at delivery. We plan to collect a breastmilk sample from the mothers in the medicated arms that have chosen to breastfeed. Clinical data related to pregnancy and neonatal health will be obtained from the prenatal and neonatal charts.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman between 18 and 40 years of age
* Have depression as their only mental health disorder
* Have been receiving fluoxetine or citalopram for the treatment of depression for at least one month on the day of study entry for patients in the fluoxetine and citalopram arms, or no pharmacological treatment for patients in the control arm
* ≤ 26 weeks pregnant by estimated date of confinement
* Ability to give informed consent
* Singleton pregnancy
* Pregnant women no history of depression

Exclusion Criteria:

* Having any comorbid mental disorder other than generalized anxiety disorder as a secondary disorder
* History of or current epilepsy, endocrine, cardiac, pulmonary, renal or hepatic dysfunction that could negatively influence pregnancy and/or neonatal outcome
* Abusing alcohol or drugs
* Use of any self prescribed herbal treatments for depression

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women up to 26 weeks gestation currently diagnosed with depression.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie L Renbarger, MD, Principal Investigator — Indiana University School of Medicine Department of Medicine and Pediatrics
Locations (1):
- IUPUI, Indianapolis, Indiana, United States